CLINICAL TRIAL: NCT06887036
Title: Methylene Blue Treatment of Chronic Hepatitis B Virus Infection: a Pilot Study
Brief Title: Methylene Blue Treatment of Chronic Hepatitis B Virus Infection
Acronym: MB_HBV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Epatocentro Ticino (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Methylene Blue in chronic HBV
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Chronic HBV Infection
Keywords: HBV; chronic HBV; Methylene Blue; MB
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Methylene Blue (Experimental): Subjects will be initially treated with an initial dose of 200mg/day for 8 weeks at which point the investigators will assess the effect of the treatment.
  Those patients that obtain a "complete response" will continue their treatment up to a total of 24 weeks with the same dose. Those who do not reach a "complete response" will be exposed to the next higher dose of 400mg/day for the following 8 weeks and the investigators will then again assess the effect of the treatment.
  Those patients that obtain a "complete response" will continue their treatment up to a total of 24 weeks with the same dose. Those who do not reach a "complete response" will be exposed to the next higher dose of 600mg/day for the following 8 weeks and the investigators will then assess the effect of the treatment.
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: Methylene Blue — Subjects will be initially treated with an initial dose of 200mg/day for 8 weeks at which point the investigators will assess the effect of the treatment.
  Those patients that obtain a "complete response" will continue their treatment up to a total of 24 weeks with the same dose. Those who do not reach a "complete response" will be exposed to the next higher dose of 400mg/day for the following 8 weeks and the investigators will then again assess the effect of the treatment.
  Those patients that obtain a "complete response" will continue their treatment up to a total of 24 weeks with the same dose. Those who do not reach a "complete response" will be exposed to the next higher dose of 600mg/day for the following 8 weeks and the investigators will then assess the effect of the treatment.

SUMMARY:
HBV infection is a global public health problem. It is estimated that there are more than 250 million HBV carriers worldwide, of whom approximately 600,000 die each year from HBV-related liver disease. Diagnosis and treatment depend on the stage of infection, the degree of liver inflammation, and the progression of fibrosis. Patients with HBeAg-positive or -negative hepatitis are usually treated with nucleos(-t)ide analogues. This treatment inhibits HBV reverse transcriptase and reduces viral replication, but does not affect HBsAg production. Treatment must be continued for life in most cases and is associated with high cumulative costs and the risk of development of resistance.

Recently, it has been shown that patients who show a decrease in their HBsAg levels are more likely to become HBsAg negative, seroconvert and be able to stop antiviral treatment, which is the ultimate goal of treatment, but unfortunately rarely achieved. Methylene blue (MB) has been shown to have an effect on HBsAg levels in vitro, making it a promising test for a new treatment for HBV.

This is an explorative pilot study, open label, dose-escalation, single center clinical trial on the efficacy of MB against HBV infection.

Primary objective is to assess the efficacy of incremental doses of MB against hepatitis B virus in patients with chronic hepatitis B assessed by the reduction of both the HBsAg and HBV DNA levels after 6 months of treatment and 6 months of follow-up.

Participant will be treated for 6 months with MB 100 mg capsules, and then followed up for a further 6 months. The initial dose of MB might be increased if the patient is a non-responder.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 and < 80 years
* Microbiologically confirmed chronic Hepatitis B Virus infection (according to the old terminology "inactive HBV carrier")
* HBsAg levels within 20-15'000 IU/ml measured at the at least twice at 6-18 months apart
* HBV DNA PCR levels within 1'000-20'000 IU/ml measured at least twice at 6-18 months apart
* Negative pregnancy test in women of child-bearing age

Exclusion Criteria:

* Documented refusal to participate in the study
* Known G-6-Phophatase deficiency
* Treatment with a serotoninergic drug
* Ongoing treatment with a nucleos(-t)ide treatment
* Clinically relevant concomitant liver disease
* GPT > 2xULN
* Fibroscan of > 8.0 KPa obtained ≤ 12 months before Visit 0/Screening
* HBeAg positivity
* Anti HDV antibody positivity
* Breastfeeding women

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Reduction >1 log10 in the starting HBsAg level and > 2 log10 in the starting HBV DNA PCR level | From enrollment to the end of treatment at 6 months
  Primary endpoints have been created according to the levels of HBsAg and HBV DNA PCR. The main primary endpoint is the reduction >1 log10 in the starting HBsAg level and > 2 log10 in the starting HBV DNA PCR level after 6 months of treatment (complete response).

SECONDARY OUTCOMES:
Adverse Events | From enrollment to the end of follow up period (12 months in total)
  Adverse Events during both the 6 months treatment period and the 6 months follow-up period after the treatment
Treatment adherence | From enrollment to the end of follow up period (12 months in total)
  Assessment of treatment adherence, through IMP accountability

CONTACTS AND LOCATIONS:
Locations (1):
- Epatocentro Ticino, Lugano, Canton Ticino, Switzerland